CLINICAL TRIAL: NCT07229625
Title: A Phase III, Randomized, Controlled, Open-Label, Multicenter Study of SHR-8068 in Combination With Adebrelimab and Platinum-Containing Chemotherapy Versus Durvalumab in Combination With Platinum-Containing Chemotherapy as First-Line Treatment for Advanced Biliary Tract Cancer (BTC)
Brief Title: A Phase III Study of SHR-8068 in Combination With Adebrelimab and Platinum-Containing Chemotherapy Versus Durvalumab in Combination With Platinum-Containing Chemotherapy as First-line Treatment for Advanced Biliary Tract Cancer (BTC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-303
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Cancer
MeSH Terms: interventions — Gemcitabine; Injections; Cisplatin; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-8068 + Adebrelimab + Cisplatin and Gemcitabine Group (Experimental)
  Interventions: Drug: SHR-8068 Injection; Drug: Adebrelimab Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Cisplatin Injection
- Durvalumab + Cisplatin and Gemcitabine Group (Active Comparator)
  Interventions: Drug: Gemcitabine Hydrochloride for Injection; Drug: Cisplatin Injection; Drug: Durvalumab Injection

INTERVENTIONS:
Drug: SHR-8068 Injection — SHR-8068 injection.
  Arms: SHR-8068 + Adebrelimab + Cisplatin and Gemcitabine Group
Drug: Adebrelimab Injection — Adebrelimab injection.
  Arms: SHR-8068 + Adebrelimab + Cisplatin and Gemcitabine Group
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine Hydrochloride for injection.
Drug: Cisplatin Injection — Cisplatin injection.
Drug: Durvalumab Injection — Durvalumab injection.
  Arms: Durvalumab + Cisplatin and Gemcitabine Group

SUMMARY:
This study is a randomized, open-label, multicenter phase III clinical trial, aiming to evaluate the efficacy and safety of SHR-8068 combined with adbelimab and platinum-based chemotherapy in contrast to varicumab combined with platinum-based chemotherapy in the first-line treatment of patients with advanced BTC.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced or recurrent/metastatic biliary adenocarcinoma that is inoperable and confirmed by histology or cytology;
2. No previous systemic anti-tumor treatment has been received;
3. At least one measurable lesion that complies with the RECIST v1.1 standard;
4. ECOG PS score: 0-1 point;
5. The expected survival period is ≥ 3 months;
6. Good organ function level;
7. Negative blood pregnancy (for women of childbearing age) and not in the lactation period, adhering to efficient contraceptive requirements;
8. Patients voluntarily joined this study and signed informed consent.

Exclusion Criteria:

1. Other pathological types of cholangiocarcinoma other than adenocarcinoma;
2. Malignant tumor of the ampulla;
3. Have had or concurrently suffered from other malignant tumors;
4. Those with concurrent biliary obstruction and at risk of biliary tract infection;
5. Those with any active or known autoimmune diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 15 months.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 7 months.
Duration of Response (DoR) | Up to 7 months.
Progression free Survival (PFS) | Up to 7 months.
Objective Response Rate (ORR) | Up to 7 months.
Time to Progression (TTP) | Up to 7 months.
Time to Response (TTR) | Up to 7 months.
Adverse events (AEs) | Up to approximately 15 months.
Serious adverse events (SAEs) | Up to approximately 15 months.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided